CLINICAL TRIAL: NCT04441203
Title: Patient SELF-management With HemodynamIc Monitoring: Virtual Heart Failure Clinic and Outcomes (the SELFIe-HF Trial): Program
Brief Title: Patient SELF-management With HemodynamIc Monitoring: Virtual Heart Failure Clinic and Outcomes
Acronym: SELFIe-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Anique Ducharme, MD, MSc. Director of the Heart Failure clinic, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHICC-2018-001
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Intervention Model Description: This will be a single center, prospective, randomized, open-label blinded-endpoint (PROBE) trial in which the treatment group will be implanted with a CardioMEMS HF sensor and managed using remote access to hemodynamics compared to a non-implanted control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Heart failure clinic follow up
- CardioMems (Active Comparator): The treatment group will be implanted with a CardioMEMS HF sensor and managed using remote access to hemodynamics compared to a non-implanted control group.
  Interventions: Device: CardioMems

INTERVENTIONS:
Device: CardioMems — novel implantable sensor inserted into the right pulmonary artery that measures pulmonary artery pressures (PAP) in patients with HF, the CardioMEMS™ HF System
  Arms: CardioMems

SUMMARY:
To demonstrate that a virtual Heart Failure Clinic (HFC) based on patient self-management using Pulmonary Artery Pressure (PAP) monitoring is superior to usual care of HFC, leads to decreased: hospital admissions for heart failure (HF), emergency department consultation and/or unplanned intravenous heart failure therapy and cardiovascular death, compared to a regular HFC, has low device-related complications and is cost-effective, in New York Heart Association (NYHA) class III and II (requiring diuretics) patients.

DETAILED DESCRIPTION:
This will be a single center, prospective, randomized, open-label blinded-endpoint (PROBE) trial in which the treatment group will be implanted with a CardioMEMS HF sensor and managed using remote access to hemodynamics compared to a non-implanted control group. Patients with at least one hospitalization for HF (≥1) in the previous year (12 months) will be randomized into two groups, regardless of LVEF:

Usual care with the specialized multidisciplinary HF clinic team (Non-implanted Control) or Hemodynamic monitoring, less intense HF clinic follow-up, and remote follow-up by a nurse clinician and patient empowerment with access to the PAP data (CardioMEMS group).

Primary and secondary endpoints will be compared between groups after 12 months of follow-up and within groups comparing baseline parameters with 12 month follow-up measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old.
2. Symptomatic HF (NYHA III) with recent heart failure admission in the previous year (12 months). OR
3. Patient with at least one ER visit or unplanned HF clinic requiring iv diuretics within 12 months will be eligible if they have in addition a N-terminal pro-BNP (NT-proBNP) level > 800pg/ml at screening AND NYHA Class II on diuretics (furosemide ≥ 40mg qd), III or ambulatory IV.
4. HF with reduced or preserved EF of at least 3 months duration.
5. Minimum technological knowledge either with a smartphone or iPAD for use of the self-management application, including access to internet.
6. Anatomical criteria

   1. PA branch diameter between 7 mm - 15 mm
   2. For BMI >35, distance from patient's back to target PA<10cm

Exclusion Criteria:

1. Recent cardiovascular event: Acute coronary syndrome (STEMI/NSTEMI; a small rise in the troponin level would be expected in this population and is not a contraindication for enrolment); Percutaneous Coronary Intervention (PCI), new cardiac rhythm management (CRM) device (pacemaker, ICD and CRT), CRM system revision, lead extraction or cardiac or other major surgery or transient ischemic attack or stroke within 2 months (3 months of stabilization after CRT or cardiac surgery);
2. Scheduled cardiac surgery;
3. History of pulmonary embolism or recurrent deep vein thrombosis;
4. Persistent NYHA Class IV and ACC/AHA HF Stage D, patients implanted with a ventricular assist device (VAD), or patients listed for cardiac transplantation and likely to be transplanted within 12 months;
5. Coexisting severe stenotic valve lesions, endocarditis, obstructive hypertrophic cardiomyopathy, acute myocarditis, tamponade, or large pericardial effusion;
6. Clinically too unstable to be followed remotely; this includes but is not limited to:

   1. Resting systolic blood pressure < 80 or > 180 mmHg;
   2. Resting heart rate > 100 bpm;
   3. Stage IV or V chronic kidney disease (Estimated Glomerular Filtration Rate (eGFR) that remains < 30 mL/min/1.73m2 by MDRD) or nonresponsive to diuretic therapy or on chronic renal dialysis;
7. Severe pulmonary hypertension with systolic pulmonary artery pressure ≥80 mmHg;
8. Pulmonary hypertension other than group II PH;
9. Anemia requiring transfusions, iron infusions, or hemoglobin below 100;
10. Coagulopathy or uninterruptible anticoagulation therapy or contraindication to antiplatelet/anticoagulant treatments anticipated in the protocol;
11. Intolerance to aspirin or clopidogrel;
12. Active infection requiring systemic antibiotics;
13. Unwillingness to sign informed consent or to attend the outpatient clinic;
14. Participation in another research trial with intervention;
15. Discharge to a chronic care facility or residence in an outlying area;
16. Pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception, such as the oral contraceptive pill, an intrauterine device or surgical sterilization. If necessary a negative urine or blood test will be performed before randomization
17. Any condition that in the opinion of the investigator would jeopardize the evaluation for efficacy or safety or be associated with poor adherence to the protocol, including cognitive decline.
18. Life expectancy <1 year;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
first occurrence of any component of the composite event | 12 months
  acute decompensated heart failure requiring emergency department consultation
Number of Participants with unplanned intravenous heart failure therapy in an outpatient clinic | 12 months
  unplanned intravenous heart failure therapy in an outpatient clinic
Number of Participants with hospital admission for heart failure | 12 months
  hospital admission for heart failure
Number of Participants with cardiovascular (CV) death | 12 months
  cardiovascular (CV) death

SECONDARY OUTCOMES:
Time to the first occurrence of the individual components of the primary endpoint | 12 months
  Acute decompensated heart failure that requires emergency department consultation and/or unplanned intravenous heart failure therapy in an outpatient clinic
Number of Participants with CV death | 12 months
  CV death
Change in Quality of life | 12 months
  Quality of life questionnaire
Change in functional capacity between baseline and 12-months | 12 months
  NYHA functional class (Kansas city cardiomyopathy questionnaire)
Change in 6 minutes walk distance | 12 months
  6 minutes walk distance test
Number of Participants with device-related endpoints | 12 months
  Safety: adverse events related to the device
Number of successful patient contacts | 12 months
  Number of successful patient contacts
Pulmonary artery pressures changes mesured by the CardioMems device | 12 months
  Pulmonary artery pressures changes mesured by the CardioMems device
Cost-effectiveness | 12 months
  cost-effectiveness ratio

CONTACTS AND LOCATIONS:
Overall Officials: Anique Ducharme, Principal Investigator — Montreal Heart Institute; Jean Rouleau, MD, Study Director — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04441203/Prot_SAP_000.pdf